CLINICAL TRIAL: NCT01323686
Title: Empiric Versus Imaging Guided Left Ventricular Lead Placement in Cardiac Resynchronization Therapy
Acronym: ImagingCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sksCRT
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imaging guided LV lead placement (Experimental)
  Interventions: Other: Imaging guided optimal LV lead placement
- Empiric LV lead placement (No Intervention): LV lead placement using standard clinical routine.

INTERVENTIONS:
Other: Imaging guided optimal LV lead placement — LV lead placement guided by cardiac imaging using echocardiography, single-photon emission computed tomography, and CT to target a cardiac vein at the site of latest mechanical activation without scar tissue.
  Visualization of cardiac venous anatomy is performed using cardiac CT if not contraindicated by depressed renal function (estimated glomerular filtration rate <30 ml/min) or allergy to contrast media. In that case, a coronary venogram is used.
  Arms: Imaging guided LV lead placement

SUMMARY:
The aim of this study is to investigate if imaging guided optimal left ventricular (LV) lead placement improves the response rate to cardiac resynchronization therapy (CRT). Consecutive patients meeting the standard criteria for CRT are included in a prospective, double-blinded, randomized trial to LV lead positioning either 1) guided by cardiac imaging using echocardiography, single-photon emission computed tomography, and visualization of cardiac venous anatomy (cardiac computed tomography (CT), venography) to target an epicardial vein at the site of latest mechanical activation without scar tissue or 2) using standard LV lead placement.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure (New York Heart Association functional class II - IV) despite stabile optimal medical therapy.
* ECG with QRS ≥ 120 milliseconds and left bundle branch block (LBBB) or paced QRS ≥ 180 milliseconds.
* LV systolic dysfunction (Ejection Fraction ≤ 35%).
* written informed consent.

Exclusion Criteria:

* Expected lifetime < 6 months.
* Recent myocardial infarction (< 3 months).
* Pregnant or lactating.
* Inadequate echocardiographic images for determination of site with latest mechanical activation
* No written informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinical response to CRT | 6 months after CRT implantation
  Response to CRT defined as a combination of survival, free of hospitalization for heart failure, and improved functional status. The primary endpoint is attained if the patient is registered for one of the following three events:
  1. Death from any cause.
  2. Hospitalization for heart failure.
  3. No improvement in New York Heart Association (NYHA) functional class and <10% improvement in 6-minutes hall walk at end of study period.

SECONDARY OUTCOMES:
All cause mortality | 6 months after CRT implantation
Hospitalization for heart failure | 6 months after CRT implantation
Changes in NYHA functional class | 6 months after CRT implantation
Changes in 6-Minutes Hall Walk | 6 months after CRT implantation
Changes in Quality of Life | 6 months after CRT implantation
  Using Minnesota Living with Heart Failure questionnaire.
Changes in Biochemical marker of heart failure | 6 months after CRT implantation
  Nt-ProBNP
Changes in LV Ejection Fraction | 6 months after CRT implantation
Changes of LV end-diastolic volume | 6 months after CRT implantation
Changes of LV end-systolic volume | 6 months after CRT implantation
Changes of LV dyssynchrony | 6 months after CRT implantation
Changes of mitral regurgitation grade | 6 months after CRT implantation
Duration of CRT implantation | During CRT implantation
Complications | 6 months after CRT implantation

CONTACTS AND LOCATIONS:
Overall Officials: Jens C. Nielsen, Professor, PhD, DMSc, Study Chair — Aarhus University Hospital; Anders Sommer, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Fyenbo DB, Norgaard BL, Blanke P, Sommer A, Duchscherer J, Kalk K, Kronborg MB, Jensen JM, McVeigh ER, Delgado V, Leipsic J, Nielsen JC. Geometric Changes in Mitral Valve Apparatus during Long-term Cardiac Resynchronization Therapy as Assessed with Cardiac CT. Radiol Cardiothorac Imaging. 2024 Oct;6(5):e230320. doi: 10.1148/ryct.230320. PMID 39360929
- [Derived] Sommer A, Kronborg MB, Poulsen SH, Bottcher M, Norgaard BL, Bouchelouche K, Mortensen PT, Gerdes C, Nielsen JC. Empiric versus imaging guided left ventricular lead placement in cardiac resynchronization therapy (ImagingCRT): study protocol for a randomized controlled trial. Trials. 2013 Apr 26;14:113. doi: 10.1186/1745-6215-14-113. PMID 23782792